CLINICAL TRIAL: NCT06579105
Title: A Phase IIb, Randomized, Double-blind, Placebo-controlled and Open-label Active Comparator Study to Evaluate the Efficacy, Safety, and Tolerability of AZD5004 in Adults With Type 2 Diabetes Mellitus.
Brief Title: Efficacy, Safety, and Tolerability of Once Daily Oral Administration of AZD5004 Versus Placebo for 26 Weeks in Adults With Type 2 Diabetes Mellitus.
Acronym: SOLSTICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D7261C00001; 2024-512562-34-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking (blinding) applies to patients and investigators involved in AZD5004 and placebo arms, however not in active comparator arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm 1 (Experimental): Participants will receive xx mg once daily dose of AZD5004
  Interventions: Drug: AZD5004
- Arm 2 (Experimental): Participants will receive xx mg once daily dose of AZD5004
  Interventions: Drug: AZD5004
- Arm 3 (Experimental): Participants will receive xx mg once daily dose of AZD5004
  Interventions: Drug: AZD5004
- Arm 4 (Experimental): Participants will receive xx mg once daily dose of AZD5004
  Interventions: Drug: AZD5004
- Arm 5 (Experimental): Participants will receive xx mg once daily dose of AZD5004
  Interventions: Drug: AZD5004
- Arm 6 (Experimental): Participants will receive xx mg once daily dose of AZD5004
  Interventions: Drug: AZD5004
- Arm 7 (Active Comparator): Participants will receive once daily dose of Semaglutide as active comparator
  Interventions: Drug: Semaglutide
- Arm 8 (Placebo Comparator): Participants will receive matching placebo for each AZD5004 arm
  Interventions: Drug: Placebo (placebo matching AZD5004 film-coated tablet)

INTERVENTIONS:
Drug: Placebo (placebo matching AZD5004 film-coated tablet) — Placebo film-coated tablet (matching AZD5004)
  Arms: Arm 8
Drug: AZD5004 — AZD5004 film-coated tablet, once daily during 26 weeks
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5; Arm 6
Drug: Semaglutide — 3-14 mg tablets of Semaglutide
  Other Names: Rybelsus
  Arms: Arm 7

SUMMARY:
This is a Phase IIb, randomised, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy, safety and tolerability of AZD5004 in adults with type 2 diabetes mellitus, compared to placebo and active comparator.

DETAILED DESCRIPTION:
This is a Phase IIb, randomised, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy, safety and tolerability of AZD5004 in adults with type 2 diabetes mellitus, compared to placebo and active comparator. The study is planned to be conducted in approximately 15 countries, approximately 90 sites will be involved.

ELIGIBILITY:
Inclusion Criteria:

Adults ≥ 18 years of age.

Diagnosed with T2DM for at least 6 months.

HbA1c ≥ 7.0% and ≤ 10.5% managed with diet and exercise alone or with a stable dose of metformin or an SGLT2 inhibitor for at least one month prior to screening.

Body mass index of ≥ 23 kg/m2.

Stable self-reported body weight for 3 months prior to randomization (+/- 5% body weight change).

Exclusion Criteria:

Type 1 diabetes mellitus, secondary forms of diabetes or history of ketoacidosis or hyperosmolar coma.

History of proliferative diabetic retinopathy, diabetic maculopathy, or severe non-proliferative diabetic retinopathy that required immediate treatment.

Have had more than one episode of severe hypoglycemia within 6 months prior to screening, or has a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms.

Received medication for weight loss within the last 3 months prior to screening.

Clinically significant inflammatory bowel disease, gastroparesis, severe disease or surgery affecting the upper GI tract.

Previous or planned (within study period) bariatric surgery or fitting of a weight loss device (eg, gastric balloon or duodenal barrier).

History of acute or chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline to Week 26
  To evaluate the effect of AZD5004 versus placebo on glycemic control

SECONDARY OUTCOMES:
Change in fasting glucose | Baseline to Weeks 4, 12, 16 and 26
  To evaluate the effect of AZD5004 versus placebo on fasting glucose
Achievement of HbA1c ≤ 6.5% | Week 26
  To evaluate of the effect of AZD5004 versus placebo on HbA1c
Baseline HbA1c ≥ 7.0% and achieved HbA1c < 7.0% | Week 26
  To evaluate the effect of AZD5004 versus placebo on HbA1c
Percent change in body weight | Baseline to Week 26
  To evaluate the effect of AZD5004 versus placebo on weight loss
Absolute change in body weight | Baseline to Week 26
  To evaluate the effect of AZD5004 versus placebo on weight loss
Achievement of ≥ 5%, ≥ 10%, and ≥ 15% weight reduction | Baseline to Week 26
  To evaluate the effect of AZD5004 versus placebo on weight loss

CONTACTS AND LOCATIONS:
Locations (91):
- United States (50):
  - Research Site, Mobile, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Vestavia Hills, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Sacramento, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Lake City, Florida
  - Research Site, Largo, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Orlando, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Lombard, Illinois
  - Research Site, Potomac, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Roslindale, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Gulfport, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Albuquerque, New Mexico
  - Research Site, Binghamton, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Beachwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Medford, Oregon
  - Research Site, West Chester, Pennsylvania
  - Research Site, Gaffney, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Abilene, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, West Jordan, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Kingwood, West Virginia
- Canada (6):
  - Research Site, Surrey, British Columbia
  - Research Site, Brampton, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
- Germany (6):
  - Research Site, Falkensee
  - Research Site, Hamburg
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Sankt Ingbert
  - Research Site, Wangen
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Matsuyama
  - Research Site, Shinjuku-ku
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Tarnów
- Slovakia (5):
  - Research Site, Bratislava
  - Research Site, Prešov
  - Research Site, Rožňava
  - Research Site, Sabinov
  - Research Site, Trebišov
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- United Kingdom (7):
  - Research Site, Blackpool
  - Research Site, Bristol
  - Research Site, Chesterfield
  - Research Site, Corby
  - Research Site, Dundee
  - Research Site, Rotherham
  - Research Site, Yate

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/